CLINICAL TRIAL: NCT01460550
Title: Comparison Between Antecolic and Retrocolic Gastrointestinal Reconstruction in Delayed Gastric Emptying After Pancreaticoduodenectomy: A Prospective Randomized Controlled Multicenter Trial
Brief Title: A Prospective Randomized Controlled Multicenter Trial of Delayed Gastric Emptying (DGE) After Pancreaticoduodenectomy Evaluating by Gastrointestinal Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Ippei Matsumoto, Associate Professor, Kobe University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KOPAS01
Record Dates: First submitted 2011-10-11; First posted 2011-10-27 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Postprocedural Delayed Gastric Emptying
Keywords: delayed gastric emptying(DGE); pancreaticoduodenectomy(PD); randomized controlled trial(RCT); gastro- or duodeno- jejunostomy reconstruction; morbidity
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gastrointestinal reconstruction (Experimental)
  Interventions: Procedure: Retrocolic gastro- or duodeno- jejunostomy in hte pancreaticoduodenectomy; Procedure: Antecolic gastro- or duodeno- jejunostomy in the pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Retrocolic gastro- or duodeno- jejunostomy in hte pancreaticoduodenectomy — The duodenojejunostomy or gastrojejunostomy was constructed in two layers or single layer. For the retrocolic reconstruction, the jejunal loop was anastomosed to the duodenum or stomach through a separate mesocolic window on the left of the middle colic vessels.
Procedure: Antecolic gastro- or duodeno- jejunostomy in the pancreaticoduodenectomy — The duodenojejunostomy or gastrojejunostomy was constructed in two layers or single layer. For the antecolic reconstruction, the jejunal loop about 30 cm distal to the hepaticojejunostomy, was brought up anterior to the transverse colon and anastomosed to the duodenum or stomach.

SUMMARY:
The purpose of this study is to evaluate the incidence of delayed gastric emptying in patient with pancreaticoduodenectomy between antecolic and retrocolic gastrointestinal reconstruction.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the incidence of delayed gastric emptying in patient with pancreaticoduodenectomy between antecolic and retrocolic gastrointestinal reconstruction. Delayed gastric emptying after pancreaticoduodenectomy is important to affect the postoperative course and QOL. We conducted a prospective randomized trial on 240 patients who underwent pancreaticoduodenectomy for comparing between antecolic and retrocolic gastrointestinal reconstruction.

The primary endpoint was defined as incidence of delayed gastric emptying by ISGPS criteria. The secondary endpoint was defined as incidence of other postoperative morbidity. Patients were recruited into this study before surgery, on the basis of whether pancreatic head resection was anticipated for pancreatic head and periampullary disease, and an appropriate informed consent was obtained. Exclusion criteria was 1) patients who have the history of gastrectomy, 2) patients who have severe cardiorespiratory dysfunction, 3) patients who have liver cirrhosis or are receiving dialysis, and 4) patients who were diagnosed inadequate for this study by a physician.

ELIGIBILITY:
Inclusion Criteria:

* patients with pancreatic-biliary disease who undergo pancreaticoduodenectomy

Exclusion Criteria:

* patients who have the history of gastrectomy
* patients who have severe cardiorespiratory dysfunction
* patients who have liver cirrhosis or are receiving dialysis
* patients who were diagnosed inadequacy for this study by a physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Incident rate of delayed gastric emptying | during hospital stay after surgery, an expected average of 3 weeks
  DGE represents the inability to return to a standard diet by the end of the first postoperative week and includes prolonged nasogastric intubation of the patient. Three different grades (A,B,and C) were defined based on the impact on the clinical course and on postoperative management by ISGPS.

CONTACTS AND LOCATIONS:
Overall Officials: Yonson Ku, MD, Study Chair — Kobe University
Locations (1):
- Kobe University, Kobe, Hyōgo, Japan

REFERENCES:
- [Background] DeOliveira ML, Winter JM, Schafer M, Cunningham SC, Cameron JL, Yeo CJ, Clavien PA. Assessment of complications after pancreatic surgery: A novel grading system applied to 633 patients undergoing pancreaticoduodenectomy. Ann Surg. 2006 Dec;244(6):931-7; discussion 937-9. doi: 10.1097/01.sla.0000246856.03918.9a. PMID 17122618
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Akizuki E, Kimura Y, Nobuoka T, Imamura M, Nagayama M, Sonoda T, Hirata K. Reconsideration of postoperative oral intake tolerance after pancreaticoduodenectomy: prospective consecutive analysis of delayed gastric emptying according to the ISGPS definition and the amount of dietary intake. Ann Surg. 2009 Jun;249(6):986-94. doi: 10.1097/SLA.0b013e3181a63c4c. PMID 19474680
- [Background] Welsch T, Borm M, Degrate L, Hinz U, Buchler MW, Wente MN. Evaluation of the International Study Group of Pancreatic Surgery definition of delayed gastric emptying after pancreatoduodenectomy in a high-volume centre. Br J Surg. 2010 Jul;97(7):1043-50. doi: 10.1002/bjs.7071. PMID 20632270
- [Background] Hayashibe A, Kameyama M, Shinbo M, Makimoto S. The surgical procedure and clinical results of subtotal stomach preserving pancreaticoduodenectomy (SSPPD) in comparison with pylorus preserving pancreaticoduodenectomy (PPPD). J Surg Oncol. 2007 Feb 1;95(2):106-9. doi: 10.1002/jso.20608. PMID 17262740
- [Background] Hashimoto Y, Traverso LW. Incidence of pancreatic anastomotic failure and delayed gastric emptying after pancreatoduodenectomy in 507 consecutive patients: use of a web-based calculator to improve homogeneity of definition. Surgery. 2010 Apr;147(4):503-15. doi: 10.1016/j.surg.2009.10.034. Epub 2009 Dec 16. PMID 20018335
- [Background] Park JS, Hwang HK, Kim JK, Cho SI, Yoon DS, Lee WJ, Chi HS. Clinical validation and risk factors for delayed gastric emptying based on the International Study Group of Pancreatic Surgery (ISGPS) Classification. Surgery. 2009 Nov;146(5):882-7. doi: 10.1016/j.surg.2009.05.012. Epub 2009 Jul 18. PMID 19744455
- [Background] Tran KT, Smeenk HG, van Eijck CH, Kazemier G, Hop WC, Greve JW, Terpstra OT, Zijlstra JA, Klinkert P, Jeekel H. Pylorus preserving pancreaticoduodenectomy versus standard Whipple procedure: a prospective, randomized, multicenter analysis of 170 patients with pancreatic and periampullary tumors. Ann Surg. 2004 Nov;240(5):738-45. doi: 10.1097/01.sla.0000143248.71964.29. PMID 15492552
- [Background] Akizuki E, Kimura Y, Nobuoka T, Imamura M, Nishidate T, Mizuguchi T, Furuhata T, Hirata K. Prospective nonrandomized comparison between pylorus-preserving and subtotal stomach-preserving pancreaticoduodenectomy from the perspectives of DGE occurrence and postoperative digestive functions. J Gastrointest Surg. 2008 Jul;12(7):1185-92. doi: 10.1007/s11605-008-0513-z. Epub 2008 Apr 22. PMID 18427904
- [Background] Murakami H, Suzuki H, Nakamura T. Pancreatic fibrosis correlates with delayed gastric emptying after pylorus-preserving pancreaticoduodenectomy with pancreaticogastrostomy. Ann Surg. 2002 Feb;235(2):240-5. doi: 10.1097/00000658-200202000-00012. PMID 11807364
- [Background] Riediger H, Makowiec F, Schareck WD, Hopt UT, Adam U. Delayed gastric emptying after pylorus-preserving pancreatoduodenectomy is strongly related to other postoperative complications. J Gastrointest Surg. 2003 Sep-Oct;7(6):758-65. doi: 10.1016/s1091-255x(03)00109-4. PMID 13129553
- [Background] Horstmann O, Markus PM, Ghadimi MB, Becker H. Pylorus preservation has no impact on delayed gastric emptying after pancreatic head resection. Pancreas. 2004 Jan;28(1):69-74. doi: 10.1097/00006676-200401000-00011. PMID 14707733
- [Background] Yeo CJ, Cameron JL, Lillemoe KD, Sohn TA, Campbell KA, Sauter PK, Coleman J, Abrams RA, Hruban RH. Pancreaticoduodenectomy with or without distal gastrectomy and extended retroperitoneal lymphadenectomy for periampullary adenocarcinoma, part 2: randomized controlled trial evaluating survival, morbidity, and mortality. Ann Surg. 2002 Sep;236(3):355-66; discussion 366-8. doi: 10.1097/00000658-200209000-00012. PMID 12192322
- [Background] Park YC, Kim SW, Jang JY, Ahn YJ, Park YH. Factors influencing delayed gastric emptying after pylorus-preserving pancreatoduodenectomy. J Am Coll Surg. 2003 Jun;196(6):859-65. doi: 10.1016/S1072-7515(03)00127-3. PMID 12788421
- [Background] Chijiiwa K, Imamura N, Ohuchida J, Hiyoshi M, Nagano M, Otani K, Kai M, Kondo K. Prospective randomized controlled study of gastric emptying assessed by (13)C-acetate breath test after pylorus-preserving pancreaticoduodenectomy: comparison between antecolic and vertical retrocolic duodenojejunostomy. J Hepatobiliary Pancreat Surg. 2009;16(1):49-55. doi: 10.1007/s00534-008-0004-3. Epub 2008 Dec 16. PMID 19083149
- [Background] Hartel M, Wente MN, Hinz U, Kleeff J, Wagner M, Muller MW, Friess H, Buchler MW. Effect of antecolic reconstruction on delayed gastric emptying after the pylorus-preserving Whipple procedure. Arch Surg. 2005 Nov;140(11):1094-9. doi: 10.1001/archsurg.140.11.1094. PMID 16301447
- [Background] Nikfarjam M, Kimchi ET, Gusani NJ, Shah SM, Sehmbey M, Shereef S, Staveley-O'Carroll KF. A reduction in delayed gastric emptying by classic pancreaticoduodenectomy with an antecolic gastrojejunal anastomosis and a retrogastric omental patch. J Gastrointest Surg. 2009 Sep;13(9):1674-82. doi: 10.1007/s11605-009-0944-1. Epub 2009 Jun 23. PMID 19548039
- [Background] Tani M, Terasawa H, Kawai M, Ina S, Hirono S, Uchiyama K, Yamaue H. Improvement of delayed gastric emptying in pylorus-preserving pancreaticoduodenectomy: results of a prospective, randomized, controlled trial. Ann Surg. 2006 Mar;243(3):316-20. doi: 10.1097/01.sla.0000201479.84934.ca. PMID 16495694
- [Derived] Toyama H, Matsumoto I, Mizumoto T, Fujita H, Tsuchida S, Kanbara Y, Kadowaki Y, Maeda H, Okano K, Fukuoka M, Takase S, Shirakawa S, Terai S, Mukubo H, Ishida J, Yamashita H, Ueno K, Tanaka M, Kido M, Ajiki T, Murakami S, Nishimura K, Fukumoto T. Influence of the Retrocolic Versus Antecolic Route for Alimentary Tract Reconstruction on Delayed Gastric Emptying After Pancreatoduodenectomy: A Multicenter, Noninferiority Randomized Controlled Trial. Ann Surg. 2021 Dec 1;274(6):935-944. doi: 10.1097/SLA.0000000000004072. PMID 32773628
- See also: Click here for more information about this study: Clinical Trial of DGE after PD — http://www.med.kobe-u.ac.jp/hbps/index.html